CLINICAL TRIAL: NCT04652193
Title: Does Obesity Effect the Recovery Profile in Children?
Brief Title: The Effect of Obesity on Recovery Profile in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Mehmet SARGIN, Associate Professor, Selcuk University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 42001
Record Dates: First submitted 2020-11-20; First posted 2020-12-03 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Recovery profile from general anesthesia — It includes the phases during recovery from general anesthesia: Time to spontaneous ventilation, Laryngeal Mask Airway (LMA) removal time, open eyes, and Post-Anesthesia Care Unit (PACU) discharge.

SUMMARY:
It is planned to investigate whether obesity affects the recovery profile after anesthesia in pediatric patients. To evaluate recovery profile, time to spontaneous ventilation (the time between anesthetic discontinuation and beginning of spontaneous ventilation), LMA removal time (the time between anesthetic discontinuation and LMA removal), open eyes (the time between anesthetic discontinuation and eye opening in response to verbal stimulus or painful pinching), and PACU discharge will be also noted.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I and II
* Routine surgery under general anesthesia

Exclusion Criteria:

* Any known cerebrovascular disease
* Long- or short-term (within the previous 24 hours) intake of any drug acting in the central nervous system
* The patients bypassing the recovery room

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Time to spontaneous ventilation | up to 20 minutes
  The time between anesthetic discontinuation and beginning of spontaneous ventilation.
LMA removal time | up to 25 minutes
  The time between anesthetic discontinuation and LMA removal.
Time to open eyes | up to 30 minutes
  The time between anesthetic discontinuation and eye opening in response to verbal stimulus or painful pinching
PACU discharge time | up to 45 minutes
  The time between entering and leaving the PACU.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University Medical Faculty Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided